CLINICAL TRIAL: NCT05785052
Title: Biomarkers of Renal Cancer
Acronym: BRC
Status: Recruiting | Type: Observational
Sponsor: Biorek S.R.L. (Industry)
Responsible Party: Sponsor
Other Study IDs: BRC
Record Dates: First submitted 2023-03-14; First posted 2023-03-27 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Renal Cell Carcinoma; Tumor, Solid; Oncocytoma; Angiomyolipoma
Keywords: Biomarkers; Urology; Renal Cell Carcinoma; Molecular Biomarkers; Oncology
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasms; Adenoma, Oxyphilic; Angiomyolipoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The samples will be fractionated and subjected to different analysis, such as the detection of nucleic acids (DNA and RNA), and proteins. These macromolecules will be purified and analyzed by employing methods such as real time PCR, microarrays, sequencing, ELISA assays, or mass spectrometry.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Renal-mass patients: Patients diagnosed with a first episode of renal mass attending the urology department.
- Control subjects: Patients affected by urological functional diseases or living kidney donor.

SUMMARY:
The aim of the present study is the identification, in liquid biopsies, of a new molecular panel able to discriminate renal cancer patients from controls, to discriminate patients with a malignant lesion from those with a benign mass, to determine aggressiveness of RCC, and to differentiate the most common histological subtypes of RCC (clear cell, papillary 1, papillary 2, and chromophobe).

This new molecular panel will be combined with clinical parameters to provide a screening test and to improve the accuracy and specificity of diagnosis, prognosis, and histological classification of renal cancer.

DETAILED DESCRIPTION:
The study is a translational one of the duration of 7 years and it is composed by a retrospective and a prospective phases.

1. Retrospective phase:

   Retrospective analysis of liquid and solid biopsies of patients diagnosed with a first episode of renal mass (of any histological subtype, such as clear cell RCC, type 1 and type 2 papillary RCC, chromophobe RCC, oncocytoma, and angiomyolipoma) and treated with radical or partial nephrectomy, in order to identify specific biomarkers for the screening, diagnosis, prognosis, and histological classification of renal cancer.

   Patients with a first episode of renal mass whose plasma, urine, tumor and matched normal kidney tissue, and PBMC have been collected and stored in a biobank since 2011, will be stratified in different groups according to (i) the nature of renal mass (benign or malignant), (ii) the aggressiveness of renal cancer (indolent kidney cancer or aggressive kidney cancer), and (iii) the presence or absence of clinical metastasis; (iv) specific histotype of renal mass (e.g., clear cell RCC, type 1 and type 2 papillary RCC, chromophobe RCC, oncocytoma, and angiomyolipoma).

   The same type of biological samples mentioned above from patients affected by urological functional diseases (such as kidney stones or benign prostate hypertrophy) have been collected and stored in a biobank between 2014 and 2018 and will be also analyzed as controls.

   The samples will be fractionated and subjected to different analysis, such as the detection of nucleic acids (DNA and RNA), and proteins. These macromolecules will be purified and analyzed by employing methods such as real time PCR, microarrays, sequencing, ELISA assays, or mass spectrometry.
2. Prospective phase and multicenter trial:

Validation of the biomarker panel in a wider cohort of patients affected by renal mass.

An ideal tumor marker is easily detected and dosed, is sensitive and specific and its clinical significance is easy to deduce. To confirm the results obtained in archived samples and validate a panel of biomarkers to be translate in the clinical practice, it will be collected whole blood, plasma and urine samples from a validation cohort of patients.

It will enrolled patients affected by renal masses (e.g., clear cell RCC, type 1 and type 2 papillary RCC, chromophobe RCC, oncocytoma, and angiomyolipoma), who will undergo radical or partial nephrectomy, and controls (patients affected by urological functional diseases, such as kidney stones or benign prostate hypertrophy) with a ratio of 2:1 in all centers included.

For each patients, clinical data will be collected, creating a dataset with the same variables used in the discovery cohort.

The aim of this prospective phase will be to confirm that the identified molecules can improve the management of patients with RCC at all the stages of clinical decision-making, in particular for the screening, diagnosis, prognosis, and histological classification of RCC.

ELIGIBILITY:
Inclusion Criteria for renal-mass patients:

* Men and women over 18 years of age
* Diagnosis of first episode of renal mass
* Caucasian race
* Signed, informed consent

Exclusion Criteria renal-mass patients:

* Any other concomitant cancer or history of active cancer in the last 5 years
* Oncological genetic syndrome
* Previous history of renal tumour
* Urothelial cancer
* End-stage renal disease on hemodialysis
* Bilateral renal cell carcinoma

Inclusion Criteria for control subjects:

* Men and women over 18 years of age
* Caucasian race
* Living kidney donor or patient with urological functional diseases (e.g. kidney stones, benign prostate hypertrophy, etc..)
* Signed, informed consent

Exclusion criteria for control subjects:

* History of active cancer in the last 5 years
* Oncological genetic syndrome
* End-stage renal disease on hemodialysis or peritoneal dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cases: patients diagnosed with a first episode of renal mass. Control subjects: living kidney donor or patient with urological functional diseases.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-06-11 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Screening | Analysis of biological samples collected before surgery
  Identification of biomarkers able to predict the presence of a renal mass, defined as a mass either benign or malignant recorded at axial imaging examination (either CT or MRI).
Diagnosis | Analysis of biological samples collected before surgery
  Identification of biomarkers able to predict the presence of a Renal Cell Carcinoma, defined as a renal malignancy
Prognosis | Analysis of biological samples collected before surgery
  Identification of biomarkers able to predict the presence of an aggressive Renal Cell Carcinoma

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Montorsi, Principal Investigator — IRCCS San Raffaele
Locations (4):
- Italy (3):
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - IRCCS San Raffaele, Milan
  - Azienda Ospedaliera Universitaria San Luigi Gonzaga, Orbassano
- Fundació Puigvert, Barcelona, Spain

REFERENCES:
- [Background] Capitanio U, Terrone C, Antonelli A, Minervini A, Volpe A, Furlan M, Matloob R, Regis F, Fiori C, Porpiglia F, Di Trapani E, Zacchero M, Serni S, Salonia A, Carini M, Simeone C, Montorsi F, Bertini R. Nephron-sparing techniques independently decrease the risk of cardiovascular events relative to radical nephrectomy in patients with a T1a-T1b renal mass and normal preoperative renal function. Eur Urol. 2015 Apr;67(4):683-9. doi: 10.1016/j.eururo.2014.09.027. Epub 2014 Oct 3. PMID 25282367
- [Background] Chanudet E, Wozniak MB, Bouaoun L, Byrnes G, Mukeriya A, Zaridze D, Brennan P, Muller DC, Scelo G. Large-scale genome-wide screening of circulating microRNAs in clear cell renal cell carcinoma reveals specific signatures in late-stage disease. Int J Cancer. 2017 Nov 1;141(9):1730-1740. doi: 10.1002/ijc.30845. Epub 2017 Jul 7. PMID 28639257
- [Background] Chow WH, Dong LM, Devesa SS. Epidemiology and risk factors for kidney cancer. Nat Rev Urol. 2010 May;7(5):245-57. doi: 10.1038/nrurol.2010.46. PMID 20448658
- [Background] Cumberbatch MG, Rota M, Catto JW, La Vecchia C. The Role of Tobacco Smoke in Bladder and Kidney Carcinogenesis: A Comparison of Exposures and Meta-analysis of Incidence and Mortality Risks. Eur Urol. 2016 Sep;70(3):458-66. doi: 10.1016/j.eururo.2015.06.042. Epub 2015 Jul 3. PMID 26149669
- [Background] Fedorko M, Stanik M, Iliev R, Redova-Lojova M, Machackova T, Svoboda M, Pacik D, Dolezel J, Slaby O. Combination of MiR-378 and MiR-210 Serum Levels Enables Sensitive Detection of Renal Cell Carcinoma. Int J Mol Sci. 2015 Sep 29;16(10):23382-9. doi: 10.3390/ijms161023382. PMID 26426010
- [Background] Gatto F, Maruzzo M, Magro C, Basso U, Nielsen J. Prognostic Value of Plasma and Urine Glycosaminoglycan Scores in Clear Cell Renal Cell Carcinoma. Front Oncol. 2016 Nov 24;6:253. doi: 10.3389/fonc.2016.00253. eCollection 2016. PMID 27933273
- [Background] Hauser S, Wulfken LM, Holdenrieder S, Moritz R, Ohlmann CH, Jung V, Becker F, Herrmann E, Walgenbach-Brunagel G, von Ruecker A, Muller SC, Ellinger J. Analysis of serum microRNAs (miR-26a-2*, miR-191, miR-337-3p and miR-378) as potential biomarkers in renal cell carcinoma. Cancer Epidemiol. 2012 Aug;36(4):391-4. doi: 10.1016/j.canep.2012.04.001. Epub 2012 Apr 26. PMID 22542158
- [Background] Heidenreich A, Ravery V; European Society of Oncological Urology. Preoperative imaging in renal cell cancer. World J Urol. 2004 Nov;22(5):307-15. doi: 10.1007/s00345-004-0411-2. Epub 2004 Jul 30. PMID 15290202
- [Background] Hollingsworth JM, Miller DC, Daignault S, Hollenbeck BK. Five-year survival after surgical treatment for kidney cancer: a population-based competing risk analysis. Cancer. 2007 May 1;109(9):1763-8. doi: 10.1002/cncr.22600. PMID 17351954
- [Background] Iwamoto H, Kanda Y, Sejima T, Osaki M, Okada F, Takenaka A. Serum miR-210 as a potential biomarker of early clear cell renal cell carcinoma. Int J Oncol. 2014 Jan;44(1):53-8. doi: 10.3892/ijo.2013.2169. Epub 2013 Nov 7. PMID 24212760
- [Background] Kutikov A, Uzzo RG. The R.E.N.A.L. nephrometry score: a comprehensive standardized system for quantitating renal tumor size, location and depth. J Urol. 2009 Sep;182(3):844-53. doi: 10.1016/j.juro.2009.05.035. Epub 2009 Jul 17. PMID 19616235
- [Background] Linehan WM, Pinto PA, Srinivasan R, Merino M, Choyke P, Choyke L, Coleman J, Toro J, Glenn G, Vocke C, Zbar B, Schmidt LS, Bottaro D, Neckers L. Identification of the genes for kidney cancer: opportunity for disease-specific targeted therapeutics. Clin Cancer Res. 2007 Jan 15;13(2 Pt 2):671s-679s. doi: 10.1158/1078-0432.CCR-06-1870. PMID 17255292
- [Background] Ljungberg B, Bensalah K, Canfield S, Dabestani S, Hofmann F, Hora M, Kuczyk MA, Lam T, Marconi L, Merseburger AS, Mulders P, Powles T, Staehler M, Volpe A, Bex A. EAU guidelines on renal cell carcinoma: 2014 update. Eur Urol. 2015 May;67(5):913-24. doi: 10.1016/j.eururo.2015.01.005. Epub 2015 Jan 21. PMID 25616710
- [Background] Morrissey JJ, Mellnick VM, Luo J, Siegel MJ, Figenshau RS, Bhayani S, Kharasch ED. Evaluation of Urine Aquaporin-1 and Perilipin-2 Concentrations as Biomarkers to Screen for Renal Cell Carcinoma: A Prospective Cohort Study. JAMA Oncol. 2015 May;1(2):204-12. doi: 10.1001/jamaoncol.2015.0213. PMID 26181025
- [Background] Morrissey JJ, Mobley J, Figenshau RS, Vetter J, Bhayani S, Kharasch ED. Urine aquaporin 1 and perilipin 2 differentiate renal carcinomas from other imaged renal masses and bladder and prostate cancer. Mayo Clin Proc. 2015 Jan;90(1):35-42. doi: 10.1016/j.mayocp.2014.10.005. PMID 25572193
- [Background] Morrissey JJ, Mobley J, Song J, Vetter J, Luo J, Bhayani S, Figenshau RS, Kharasch ED. Urinary concentrations of aquaporin-1 and perilipin-2 in patients with renal cell carcinoma correlate with tumor size and stage but not grade. Urology. 2014 Jan;83(1):256.e9-14. doi: 10.1016/j.urology.2013.09.026. Epub 2013 Nov 13. PMID 24239027
- [Background] Pantuck AJ, Zisman A, Belldegrun AS. The changing natural history of renal cell carcinoma. J Urol. 2001 Nov;166(5):1611-23. PMID 11586189
- [Background] Redova M, Poprach A, Nekvindova J, Iliev R, Radova L, Lakomy R, Svoboda M, Vyzula R, Slaby O. Circulating miR-378 and miR-451 in serum are potential biomarkers for renal cell carcinoma. J Transl Med. 2012 Mar 22;10:55. doi: 10.1186/1479-5876-10-55. PMID 22440013
- [Background] Richard PO, Jewett MA, Bhatt JR, Kachura JR, Evans AJ, Zlotta AR, Hermanns T, Juvet T, Finelli A. Renal Tumor Biopsy for Small Renal Masses: A Single-center 13-year Experience. Eur Urol. 2015 Dec;68(6):1007-13. doi: 10.1016/j.eururo.2015.04.004. Epub 2015 Apr 18. PMID 25900781
- [Background] Siegel R, Naishadham D, Jemal A. Cancer statistics, 2012. CA Cancer J Clin. 2012 Jan-Feb;62(1):10-29. doi: 10.3322/caac.20138. Epub 2012 Jan 4. PMID 22237781
- [Background] Teixeira AL, Ferreira M, Silva J, Gomes M, Dias F, Santos JI, Mauricio J, Lobo F, Medeiros R. Higher circulating expression levels of miR-221 associated with poor overall survival in renal cell carcinoma patients. Tumour Biol. 2014 May;35(5):4057-66. doi: 10.1007/s13277-013-1531-3. Epub 2013 Dec 31. PMID 24379138
- [Background] Thompson RH, Ordonez MA, Iasonos A, Secin FP, Guillonneau B, Russo P, Touijer K. Renal cell carcinoma in young and old patients--is there a difference? J Urol. 2008 Oct;180(4):1262-6; discussion 1266. doi: 10.1016/j.juro.2008.06.037. Epub 2008 Aug 15. PMID 18707708
- [Background] Wang C, Hu J, Lu M, Gu H, Zhou X, Chen X, Zen K, Zhang CY, Zhang T, Ge J, Wang J, Zhang C. A panel of five serum miRNAs as a potential diagnostic tool for early-stage renal cell carcinoma. Sci Rep. 2015 Jan 5;5:7610. doi: 10.1038/srep07610. PMID 25556603
- [Background] Wulfken LM, Moritz R, Ohlmann C, Holdenrieder S, Jung V, Becker F, Herrmann E, Walgenbach-Brunagel G, von Ruecker A, Muller SC, Ellinger J. MicroRNAs in renal cell carcinoma: diagnostic implications of serum miR-1233 levels. PLoS One. 2011;6(9):e25787. doi: 10.1371/journal.pone.0025787. Epub 2011 Sep 30. PMID 21984948
- [Result] Brookman-May SD, May M, Wolff I, Zigeuner R, Hutterer GC, Cindolo L, Schips L, De Cobelli O, Rocco B, De Nunzio C, Tubaro A, Coman I, Truss M, Dalpiaz O, Feciche B, Figenshau RS, Madison K, Sanchez-Chapado M, Santiago Martin Mdel C, Salzano L, Lotrecchiano G, Zastrow S, Wirth M, Sountoulides P, Shariat S, Waidelich R, Stief C, Gunia S; CORONA Project; European Association of Urology (EAU) Young Academic Urologists (YAU) Renal Cancer Group. Evaluation of the prognostic significance of perirenal fat invasion and tumor size in patients with pT1-pT3a localized renal cell carcinoma in a comprehensive multicenter study of the CORONA project. Can we improve prognostic discrimination for patients with stage pT3a tumors? Eur Urol. 2015 May;67(5):943-51. doi: 10.1016/j.eururo.2014.11.055. Epub 2015 Feb 13. PMID 25684695